CLINICAL TRIAL: NCT03866694
Title: Growing Together: A Pragmatic Clinical Trial of a Parenting Intervention for Women in Opioid Treatment and Their Infants
Brief Title: Growing Together: Women in Opioid Treatment and Their Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency); Institute for Health and Recovery (IHR) (Unknown); Boston University (Other)
Responsible Party: Principal Investigator, Ruth Paris, Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R40MC31764
Record Dates: First submitted 2018-11-20; First posted 2019-03-07 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Substance-Related Disorders
Keywords: maternal opioid use; substance use; parent-child relationship; parenting; social and emotional development; mental health and well-being; perinatal; postpartum; health disparities
MeSH Terms: conditions — Substance-Related Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants in this randomized controlled trial are assigned to one of two groups, BRIGHT or STAR. BRIGHT is a therapeutic parenting intervention that begins in the third trimester of pregnancy and continues through six months postpartum. BRIGHT and STAR receive the standard of care at a high risk maternal-fetal medical clinic and 7 psycho-educational handouts over the course of the study.
Masking Description: No masking is used in this clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRIGHT (Experimental): Building Resilience through Intervention: Growing Healthier Together (BRIGHT) weekly home-based intervention from the third trimester of pregnancy through 6 months postpartum. A licensed clinician meets with mother and infant to promote attunement and optimal parent-child interactions. Additionally, the mother receives monthly handouts focused on information about child development and recovery from substance misuse while parenting, along with the standard of care at a high risk maternal-fetal medical clinic
  Interventions: Behavioral: BRIGHT
- STAR/TAU+ (Active Comparator): The mother receives monthly handouts focused on information about child development and recovery from substance misuse while parenting, along with the standard of care at a high risk maternal-fetal medical clinic.
  Interventions: Other: STAR/TAU+

INTERVENTIONS:
Behavioral: BRIGHT — Dyadic therapeutic parenting intervention (BRIGHT) beginning in third trimester of pregnancy through six months postpartum focusing on child-parent relationship, mental health, infant social-emotional development, and recovery. Monthly handouts for mothers in recovery with information about child development and recovery from substance misuse while parenting and the standard of care at participant's high risk maternal-fetal medical clinic.
  Arms: BRIGHT
Other: STAR/TAU+ — Monthly handouts for mothers in recovery with information about child development and recovery from substance misuse while parenting and the standard of care at participant's high risk maternal-fetal medical clinic
  Arms: STAR/TAU+

SUMMARY:
This study evaluates the effectiveness of the home-based therapeutic parenting intervention BRIGHT with pregnant women and postpartum mothers with opioid use disorders (OUDs) and their infants. It examines whether participation in the BRIGHT intervention improves parent-child relationships, parenting capacities, the mother's overall mental health, participation in OUD treatment, infant social-emotional development and decreases the likelihood of child maltreatment. Approximately half of the participants will receive the BRIGHT intervention, monthly handouts, and the standard of care at the maternal-fetal medical clinic and the other half will receive STAR, or Enhanced Treatment as Usual (TAU+), which includes monthly handouts and the standard of care from the medical clinic.

DETAILED DESCRIPTION:
Growing Together is a two-armed pragmatic randomized controlled trial of a trauma and evidence-informed therapeutic parenting intervention, BRIGHT. This trial lasts approximately 9 months.

BRIGHT has been offered to young children ages birth through 6 years and their parents affected by substance use disorders (SUDs) to mitigate the effects of trauma, promote resilience, and enhance the quality of parent-child relationships and parenting skills. BRIGHT has been successfully piloted and evaluated within residential treatment and outpatient opioid treatment programs for pregnant women/mothers with SUDs and OUDs with young children .

For this study, BRIGHT has been adapted for home-based delivery for pregnant women receiving treatment for OUDs and is offered from the 3rd trimester of pregnancy until the infant is about 6 months old. Participants in both arms will be recruited from a high-risk maternal-fetal medicine clinic and followed for approximately 15 months. The two arms of the trial are 1) the BRIGHT (Building Resilience through Intervention, Growing Healthier Together) intervention, and 2) STAR. Both arms of the study will receive the typical standard of care of at a high-risk maternal-fetal medical clinic and 7 monthly psycho-educational handouts on child development specifically for mothers in recovery.

The investigators are testing the effectiveness of the adapted version of BRIGHT by utilizing measures to examine if participation in BRIGHT decreases the likelihood of child maltreatment, improves parent-child relationships, parenting capacities, the mother's overall mental health, participation in OUD treatment, and infant social-emotional development.

ELIGIBILITY:
Inclusion Criteria:

* A patient at BUMC RESPECT clinic with history of opioid use or history of polysubstance use
* 18 years orolder
* Being treated with methadone, naltrexone, or suboxone
* In 3rd trimester of pregnancy
* Deemed by MDs able to give informed consent
* Planning to parent infant after birth
* Willing to participate in RCT

Exclusion Criteria:

* Planning to relinquish custody of neonate
* Residing, or expected to reside post-birth 20+ miles from Boston
* Deemed by MDs unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-13 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Coding Interactive Behavior (CIB) system (Observer-rated parent-infant video), measuring Maternal Sensitivity (representing the parent-child relationship) | t1 (6-8 Weeks postpartum), t2 (6-8 months postpartum)
  CIB is a rating of mother-child interactions which has three 5-point Likert subscales: Maternal Sensitivity (MSense, primary outcome), Maternal intrusiveness (MIntrude), and Child involvement. (CInvolve). High scores on CIB scales indicate more evidence of the behavior/dimension. Moderate scores typically indicate presence of the behavior/dimension approximately 50% of the time. Low scores indicate that the behavior/dimension is never/infrequently observed. The CIB has been validated with healthy and at-risk populations. The study is assessing the change in CIB score between the time points.
The Adult- Adolescent Parenting Inventory-2 (AAPI), measuring the Risk of Child Maltreatment | t1 (6-8 weeks postpartum), t2 (6-8 months postpartum), t3 (9-11 months postpartum)
  Responses to the inventory provide an index of risk for practicing behaviors known to be attributable to child abuse and neglect. Answers are recorded on a scale from Strongly Agree to Strongly Disagree. Subscales include: Construct A - Inappropriate Expectations of Children, Construct B - Parental Lack of Empathy Towards Children's Needs, Construct C - Strong Parental Belief in the Use of Corporal Punishment, Construct D - Reversing Parent-Child Family Roles, Construct E - Oppressing Children's Power and Independence. 32-item inventory assessing parenting and child-rearing attitudes associated with risk for child maltreatment. Five parenting interaction constructs include, 1) inappropriate expectations for child, 2) empathic awareness of child's needs, 3) belief in corporal punishment, 4) role reversal and 5) oppressing children's power. Construct validity is well-established. Test-re-test reliability is .76. The study is assessing the change in AAPI score between the time points.

SECONDARY OUTCOMES:
Karitane Parenting Confidence Scale (KPCS), measuring Parenting Capacity | t1 (6-8 weeks postpartum), t2 (6-8 months postpartum), t3 (9-11 months postpartum)
  15-item self-report measure of perceived parental self-efficacy, for parents of infants birth-12 months .82 The KPCS has good internal validity and test-re-test reliability is .88. Each item on the KPCS is scored 0, 1, 2, or 3, with scores summed to produce a total score. The general rule is that a high score indicates the parent is feeling confident on that item.
Parenting Stress Index/Short Form (PSI/SF), measuring Parenting Capacity | t1 (6-8 weeks postpartum), t2 (6-8 months postpartum), t3 (9-11 months postpartum)
  36-item self-report measure of parenting stress in 3 domains: parental distress, parent-child dysfunctional interaction, and parent's perceptions of child's difficulty. A high total stress score (above 90) indicates a greater level of parenting stress. The PSI/SF has excellent external validity, and test-re-test reliability is .76. Screening and triage measure for evaluating the parenting system and identifying issues that may lead to problems in the child's or parent's behavior. Focuses on three major domains of stress: child characteristics, parent characteristics and situational/demographic life stress. 1-5 Likert scale. 3 subscales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. Child and Parent domains combine to form Total Stress Scale.
The Parental Reflective Functioning Questionnaire (PRFQ), measuring Parenting Capacity | t1 (6-8 weeks postpartum), t2 (6-8 months postpartum), t3 (9-11 months postpartum)
  Multidimensional assessment of parental reflective functioning in parents with children 0-5 years old. 1-7 Likert scale (1= Strongly Disagree, 7= Strongly Agree). 39-item measure of levels of reflective functioning - parent's ability to reflect upon and "see" their child's internal experiences, including wishes, fears, intentions, and emotions that drive children's behavior. Higher levels of reflective functioning indicate abilities to respond in a more empathetic and supportive manner. The PRFQ has good internal consistency and discriminant validity.
The Brief Symptom Inventory (BSI), measuring Maternal Mental Health (including continuation of OUD treatment) | t0 (3rd trimester), t1 (6-8 weeks postpartum), t2 (6-8 months postpartum)
  Provides an overview of a patient's psychological symptoms and their intensity at a specific point in time. 0-4 Likert scale, lower scores are "better." 53-item self-report measure of mothers' psychological distress. Dimensions include depression, somatization, obsession-compulsion, anxiety, hostility, phobic anxiety, interpersonal sensitivity, paranoid ideation, and psychoticism. The BSI is known to have good reliability and validity.
The Life Stressor Checklist- Revised (LSC-R), measuring Maternal Mental Health (including continuation of OUD treatment) | t0 (3rd trimester)
  22-item, self-report measure of traumatic or stressful life events. Stressful events are rated for occurrence (yes/no) and the age(s) of occurrence. The LSC-R maintains good criterion validity and test-retest reliability. A lower score is "better."
Connor-Davidson Resilience Scale-10 (CD-RISC 10), measuring Maternal Mental Health (including continuation of OUD treatment) | t0 (3rd trimester), t1 (6-8 weeks postpartum), t2 (6-8 months postpartum)
  10-item assessment of resilience, specifically hardiness and persistence, has demonstrated strong psychometric properties. CDRS measures "bounce-back" and adaptability in relationship to stress. 0-4 Likert scale (0= Not true at all; 4= True nearly all the time). Higher scores are considered "better."
Post Traumatic Stress Disorder Checklist (PCL-5), measuring Maternal Mental Health (including continuation of OUD treatment) | t0 (3rd trimester), t1 (6-8 weeks postpartum), t2 (6-8 months postpartum)
  20-item self-report questionnaire, corresponds to DSM-5 symptom criteria for PTSD. Rating scales span 0-4 for each symptom. The wording of PCL-5 items reflects both changes to existing symptoms and the addition of new symptoms in DSM-5. Preliminary validation work suggests a cut point of 38. 0-4 Likert scale (0= Not at all; 4= Extremely) Lower scores are considered "better."
Addiction Severity Index (ASI), measuring Maternal Mental Health (including continuation of OUD treatment) | t0 (3rd trimester), t1 (6-8 weeks postpartum), t2 (6-8 months postpartum)
  Semi-structured interview designed to address misuse of alcohol and drugs in the past 30 days and lifetime use in days and years. Lower numbers are considered "better."
Devereaux Early Childhood Assessment for Infants and Toddlers (DECA-I/T), measuring Infant Social-Emotional Development | t1 (6-8 weeks postpartum), t2 (6-8 months postpartum), t3 (9-11 months postpartum)
  Standardized assessment of protective factors and screens for social/emotional risks and development in very young children, has demonstrated very good reliability and validity.89 Parents report perceptions of their child's qualities/abilities, yielding 2 scales: infant initiative and attachment, with an overall protective factors scale. It is recommended as a research tool to assess infants' and toddlers' social-emotional outcomes. 0-4 Likert scale (0= Never, 4= Very Frequently), higher values represent better outcomes
Parent Development Interview (PDI)- Short Form Revised 2016, measuring Parental Reflective Functioning | t0 (3rd trimester), t2 (6-8 months postpartum)
  A semi-structured clinical interview that asks parents to describe the child, their internal experience of parenting, and their experience of the relationship with the child. The PI is coded by a trained and reliable PI coder using the Reflective Functioning Scale. -1 through 9 scale (-1: Negative; 9: Full or Exceptional). Higher scores indicate a high level of reflective functioning sophistication.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Paris, PhD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No